CLINICAL TRIAL: NCT03871647
Title: Effect of Genetic Polymorphism on the Occurrence of Post-Operative Atrial Fibrillation After Coronory Artery Bypass Grafting (CABG) Surgery in Egyptian Patients Receiving Beta Blockers
Brief Title: Effect of Genetic Polymorphism on the Occurrence of Post-Operative Atrial Fibrillation After CABG
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Dina Mohamed Kamal El gindy, Assistant Lecturer of Clinical Pharmacy, Misr International University
Other Study IDs: PhD 53
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Coronary Bypass Graft Surgery; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAF group: Patients who will experience AF at any time during the first six days after the operation.
  Interventions: Drug: Beta blocker
- Non POAF group: Patients with a sinus rhythm during the first six days after the operation.
  Interventions: Drug: Beta blocker

INTERVENTIONS:
Drug: Beta blocker — perioperative beta blockers

SUMMARY:
Postoperative Atrial Fibrillation (POAF) is one of the most common complications following coronary artery bypass grafting (CABG) occurring to 20% - 40% of patients. It is associated with prolonged hospitalization, increased hospital costs, increased complications and mortality rate.

Despite the use of Beta Blockers, approximately 20% of patients develop atrial fibrillation following CABG surgery, suggesting a role for polymorphism in the genes The aim of the present study is to determine the minor allele frequency of some of the genes that affect the beta blockers' response and to determine the association between polymorphism in these genes and the occurrence of postoperative atrial fibrillation after coronary artery bypass grafting in Egyptian patients receiving perioperative beta blockers.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Candidates for CABG surgery without a concurrent valve surgery.
3. Patients receiving perioperative beta blockers before new onset of postoperative AF.

Exclusion Criteria:

1. Patients who have either persistent or permanent AF, atrial flutter or atrial tachycardia on ECG obtained on the day of the operation.
2. Serum creatinine >2 mg/dL before the surgery.
3. Uncontrolled thyroid disease.
4. Recent treatment with amiodarone before the occurrence of POAF

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptian patients undergoing Coronary Artery Bypass grafting Surgery
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of Atrial fibrillation | within 6 days after the operation
  Atrial fibrillation based on postoperative electrocardiogram. AF diagnostic criteria will include absence of discrete P waves, the RR intervals follow unrepetitive form and the ranges of ventricular rate usually between 90 and 170 beats/min.

CONTACTS AND LOCATIONS:
Overall Officials: Dina M El Gindy, MSC, Principal Investigator — Misr Ineternational University; Lamiaa M ElWakeel, PhD, Study Chair — Ain Shams University; Mona F Schaalan, PhD, Study Director — Misr International University; Ramy MR Khorshid, Md, PhD, Study Director — Ain Shams Uiversity; Mohamed H Solayman, PhD, Study Director — Ain Sham University
Locations (1):
- The Cardiovascular & Thoracic Academy - Ain Shams University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El Gindy DMK, Solayman MH, Khorshid R, Schaalan MF, El Wakeel LM. Effect of Clinical and Genetic Factors on the Development of Postoperative Atrial Fibrillation After Coronary Artery Bypass Grafting (CABG) in Egyptian Patients Receiving Beta-Blockers. Cardiovasc Drugs Ther. 2024 Feb;38(1):99-108. doi: 10.1007/s10557-022-07380-6. Epub 2022 Sep 15. PMID 36107363